CLINICAL TRIAL: NCT01508182
Title: A Single-Dose, Open-Label, Randomized, 2-Way Crossover Pivotal Study to Assess the Bioequivalence of 2 FDC Tablets of Canagliflozin and Metformin IR (150 mg/500 mg) With Respect to the Individual Components of Canagliflozin (1x300 mg) and Metformin IR Tablets (2x500 mg) in Healthy Fed Subjects
Brief Title: A Study of Canagliflozin and Metformin Immediate Release (150 mg/500 mg) FDC Tablets in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100679; 28431754DIA1050 (Other: Janssen Research & Development)
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Healthy Volunteers; Bioequivalence; Canagliflozin (JNJ-28431754); Metformin IR
MeSH Terms: interventions — Canagliflozin

ARMS (2):
- Treatment Sequence AB (Experimental): Treatment A (canaglifozin + metformin IR tablets) administered on Day 1 of Treatment Period 1 followed by Treatment B (canagliflozin/metformin IR FDC tablets) administered on Day 1 of Treatment Period 2 with a washout period of 10-15 days between Treatment Periods.
  Interventions: Drug: Canagliflozin tablets; Drug: Metformin IR tablets; Drug: Canagliflozin/metformin IR FDC tablets
- Treatment Sequence BA (Experimental): Treatment B (canagliflozin/metformin IR FDC tablets) administered on Day 1 of Treatment Period 1 followed by Treatment A (canaglifozin + metformin IR tablets) administered on Day 1 of Treatment Period 2 with a washout period of 10-15 days between Treatment Periods.
  Interventions: Drug: Canagliflozin tablets; Drug: Metformin IR tablets; Drug: Canagliflozin/metformin IR FDC tablets

INTERVENTIONS:
Drug: Canagliflozin tablets — Type = exact number, unit = mg, number = 300, form = tablet, route = oral use. One canagliflozin tablet taken orally (by mouth) on Day 1 of Treatment Period 1.
  Other Names: Treatment A (Reference)
  Arms: Treatment Sequence AB
Drug: Metformin IR tablets — Type = exact number, unit = mg, number = 500, form = tablet, route = oral use. Two metformin IR tablets taken orally (by mouth) on Day 1 of Treatment Period 1.
  Other Names: Treatment A (Reference)
  Arms: Treatment Sequence AB
Drug: Canagliflozin/metformin IR FDC tablets — Type = exact number, unit = mg, number = 50/500, form = tablet, route = oral use. Two Canagliflozin/metformin IR FDC tablets taken orally on Day 1 of Treatment Period 2.
  Other Names: Treatment B (Test)
  Arms: Treatment Sequence AB
Drug: Canagliflozin tablets — Type = exact number, unit = mg, number = 300, form = tablet, route = oral use. One canagliflozin tablet taken orally (by mouth) on Day 1 of Treatment Period 2.
  Other Names: Treatment A (Reference)
  Arms: Treatment Sequence BA
Drug: Metformin IR tablets — Type = exact number, unit = mg, number = 500, form = tablet, route = oral use. Two metformin IR tablets taken orally (by mouth) on Day 1 of Treatment Period 2.
  Other Names: Treatment A (Reference)
  Arms: Treatment Sequence BA
Drug: Canagliflozin/metformin IR FDC tablets — Type = 2, unit = mg, number = 50/500, form = tablet, route = oral use. Two Canagliflozin/metformin IR FDC tablets taken orally on Day 1 of Treatment Period 1.
  Other Names: Treatment B (Test)
  Arms: Treatment Sequence BA

SUMMARY:
The purpose of this study is to evaluate the bioequivalence of fixed dose combination (FDC) tablets of canagliflozin and metformin immediate release (IR) in comparison with the individual components of the FDC tablets (canagliflozin and metformin IR).

DETAILED DESCRIPTION:
This is an open-label (identity of study drug will be known to volunteer and study staff), single-center study to evaluate the bioequivalence (to see if blood levels of one drug are equivalent to blood levels of another drug) of canagliflozin and metformin IR when administered orally (by mouth) as individual components (ie, separate tablets of canagliflozin and metformin IR) (Treatment A) and when administered as FDC tablets (ie, canagliflozin and metformin IR contained in the same tablet) (Treatment B). Healthy volunteers participating in the study will be randomly (by chance) assigned to receive a single dose of Treatment A followed by a single dose of Treatment B or Treatment B followed by Treatment A with a period of approximately 15 days between treatments. The total duration of the study will be approximately 51 days.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 and 30 kg/m² (inclusive) and a body weight of not less than 50 kg

Exclusion Criteria:

- History of or current medical illness, abnormal values for hematology or clinical chemistry laboratory tests, or abnormal physical examination, vital signs or 12-lead electrocardiogram (ECG) deemed to be clinically significant by the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Canagliflozin plasma concentrations | Up to 72 hours in Treatment Period 1 and Treatment Period 2
Metformin plasma concentrations | Up to 24 hours in Treatment Period 1 and Treatment Period 2

SECONDARY OUTCOMES:
Changes in clinical laboratory test values | Up to approximately 51 days (includes from time of screening through study completion including the washout interval)
Changes in vital signs measurements | Up to approximately 51 days (includes from time of screening through study completion including the washout interval)
Changes in electrocardiogram (ECG) parameters | Up to approximately 51 days (includes from time of screening through study completion including the washout interval)
Changes in physical examination results | Up to approximately 51 days (includes from time of screening through study completion including the washout interval)
The number of patients reporting adverse events | Up to approximately 51 days (includes from time of screening through study completion including the washout interval)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC L.L.C Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Tempe, Arizona, United States